CLINICAL TRIAL: NCT00703404
Title: A Cohort Observational Study to Assess the Virologic Response to Standard HIV Treatment in Bamako, Mali
Brief Title: Response to Standard HIV Treatment in Bamako, Mali
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999908160; 08-I-N160
Record Dates: First submitted 2008-06-20; First posted 2008-06-23 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2016-02-24

CONDITIONS: HIV Infections
Keywords: Anti-Retroviral Therapy; HIV; Virologic Response; Treatment Naïve
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This study will evaluate the effectiveness of first-line HIV treatment (fixed-dose combination of the generic antiretroviral drugs nevirapine, stavudine and lamivudine) provided by the Malian National HIV Treatment Program. Antiretroviral therapy has become a priority because of its proven effectiveness in decreasing sickness and death from HIV infection. Reliable information on its efficacy is needed.

Patients 18 years of age and older who enter the Malian National HIV Treatment Program and have not had prior antiretroviral treatment may be eligible for this study.

Primary Objective

The primary objective is to measure the virologic treatment response at 24 weeks to the Malian-approved fixed-dose regimen (FDC) of nevirapine, stavudine and lamivudine (Triomune) in patients who are na(SqrRoot) ve to antiretroviral therapy in Bamako, Mali compared to a historical cohort as a prelude to further clinical research investigations in Mali.

Secondary Objectives

1. To assess the association of the 24 week response with the response at one year as measured by suppression of viremia to less than 50 copies/mL
2. To evaluate the baseline clinical and HIV-associated characteristics of a cohort of persons who are enrolled in protocol-mandated monitoring.

Participants undergo treatment in the government-sponsored program. Clinical visits are scheduled at study days 0 (antiviral therapy start day) and 14, and at 1, 3, 6, 9 and 12 months. Patients undergo a medical history, including all confirmed and probably diagnoses made since the previous visit and current status, physical examination and blood tests for CD4 and viral load at each visit.

Study start date: July 2008

DETAILED DESCRIPTION:
This study will assess the efficacy of HIV treatment provided in accordance with the Malian National HIV Treatment Program. The Malian National HIV Treatment Program uses fixe dose coninaison (FDC) therapy, and this study will use a historical comparison from an African country in which the same generic antiretoviral are used. Virologic responses of patients enrolled in the Malian national program will be determined and, in a non-inferiority design, compared to these historical controls. The study will also establish the feasibility of doing frequent HIV virologic monitoring in this setting.

Viral RNA and CD4 T-cell count monitoring will be performed for HIV-infected persons seen at study sites. All clinical decision-making and prescription will occur outside of the protocol. Decisions about whether antiretroviral therapy is appropriate, the prescription of antiretroviral therapy, and the monitoring of treatment will be done by Malian health-care providers outside of the scope of the protocol. Viral RNA monitoring will be used to assess the endpoint of viral RNA suppression below the limit of detection (50 copies/mL).

ELIGIBILITY:
* INCLUSION CRITERIA:

HIV-infected adults (age greater than or equal to 18 years) naive to treatment with antiretroviral medications, who are to begin the regimen of government-sponsored antiretroviral treatment program or an alternate regimen in the case of HIV1 and HIV2 coinfected individuals.

The sole exception to naive will be a history of use of peripartum single-dose nevirapine.

Hemoglobin greater than or equal to 8 g/dL

Ability and willingness to provide informed consent and ability to comply with study requirements and visit schedule.

Must be willing to allow stored samples to be used in the future for studying HIV disease and immune function.

EXCLUSION CRITERIA:

Serologic evidence of HIV-2 infection mono-infection.

Tuberculosis of any form for which the patient is currently undergoing treatment with or requires a recommended regimen containing a rifamycin antibiotic.

Baseline medical conditions that preclude the use of the Malian fixed-dose regimen, such as peripheral neuropathy of any etiology and pancreatic disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2008-06-18; Study Completion 2016-02-24

CONTACTS AND LOCATIONS:
Overall Officials: Sophia B Siddiqui, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- University of Bamako, Faculty of Medicine, Pharmacy and Odontostomatology, Bamako, Mali

REFERENCES:
- [Background] Demeter LM, Hughes MD, Coombs RW, Jackson JB, Grimes JM, Bosch RJ, Fiscus SA, Spector SA, Squires KE, Fischl MA, Hammer SM. Predictors of virologic and clinical outcomes in HIV-1-infected patients receiving concurrent treatment with indinavir, zidovudine, and lamivudine. AIDS Clinical Trials Group Protocol 320. Ann Intern Med. 2001 Dec 4;135(11):954-64. doi: 10.7326/0003-4819-135-11-200112040-00007. PMID 11730396
- [Background] Anekthananon T, Ratanasuwan W, Techasathit W, Sonjai A, Suwanagool S. Safety and efficacy of a simplified fixed-dose combination of stavudine, lamivudine and nevirapine (GPO-VIR) for the treatment of advanced HIV-infected patients: a 24-week study. J Med Assoc Thai. 2004 Jul;87(7):760-7. PMID 15521230
- [Background] Idigbe EO, Adewole TA, Eisen G, Kanki P, Odunukwe NN, Onwujekwe DI, Audu RA, Araoyinbo ID, Onyewuche JI, Salu OB, Adedoyin JA, Musa AZ. Management of HIV-1 infection with a combination of nevirapine, stavudine, and lamivudine: a preliminary report on the Nigerian antiretroviral program. J Acquir Immune Defic Syndr. 2005 Sep 1;40(1):65-9. doi: 10.1097/01.qai.0000159516.39982.1b. PMID 16123684